CLINICAL TRIAL: NCT01827891
Title: Remote Ischemic Preconditioning and Risk of Contrast-Induced Acute Kidney Injury in Patients Undergoing Coronary Stent Implantation
Acronym: REPAIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, professor of cardiology, Vice president of Beijing Anzhen Hospital, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AZ-12
Record Dates: First submitted 2013-03-31; First posted 2013-04-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; percutaneous coronary intervention; remote ischemic preconditioning
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Placebo Comparator): Control participants did not experience the procedure of transient upper-limb ischemia.
- remote ischemic preconditioning (RIPC) group (Active Comparator): Those randomized to RIPC group had a pneumatic medical tourniquet cuff (width , 5 cm ; length , 40 cm) placed around their upper arm at < 2 hours before the PCI procedure. The pneumatic medical cuff was inflated to a pressure of 200 mm Hg for 5 minutes , followed by 5 minutes of deflation to allow reperfusion. This procedure was repeated for 3 times.
  Interventions: Procedure: remote ischemic preconditioning (RIPC)

INTERVENTIONS:
Procedure: remote ischemic preconditioning (RIPC) — Those randomized to RIPC group had a pneumatic medical tourniquet cuff (width , 5 cm ; length , 40 cm) placed around their upper arm at < 2 hours before the PCI procedure. The pneumatic medical cuff was inflated to a pressure of 200 mm Hg for 5 minutes , followed by 5 minutes of deflation to allow reperfusion. This procedure was repeated for 3 times.
  Arms: remote ischemic preconditioning (RIPC) group

SUMMARY:
This single-center, randomized controlled trial is to investigate the impact of remote ischemic preconditioning (RIPC) on the risk contrast-induced acute kidney injury and its long-term impact on renal function for patients with diabetes undergoing percutaneous coronary intervention.

DETAILED DESCRIPTION:
Patients with diabetes undergoing elective percutaneous coronary intervention in Beijing Anzhen Hospital were enrolled, and all the eligible participants were randomized to either remote ischemic preconditioning (RIPC) group or control group. Those randomized to RIPC group had a pneumatic medical tourniquet cuff (width , 5 cm ; length , 40 cm) placed around their upper arm at < 2 hours before the PCI procedure. The pneumatic medical cuff was inflated to a pressure of 200 mm Hg for 5 minutes , followed by 5 minutes of deflation to allow reperfusion. This procedure was repeated for 3 times. Control participants did not experience this procedure of transient upper-limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes undergoing percutaneous coronary intervention were included.

Exclusion Criteria:

1. emergency PCI,
2. baseline troponin value > 0.04 ng/mL,
3. nicorandil or glibenclamide use (preconditioning-mimetic and preconditioning-blocking medication, respectively),
4. patient on dialysis,
5. patients who had some inability to cooperate with the trial,
6. those who could not give informed consent, and (7) second procedure of staged elective PCI in this hospitalization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury | 72 hours after procedure
  The primary study endpoint was AKI, defined as an absolute rise in serum creatinine of ≥ 0.5 mg/dl or a relative increase of ≥ 25% compared to baseline within 72 hours from PCI (the maximal measured concentration of serum creatinine during these 72 hours was used).

SECONDARY OUTCOMES:
relative reduction in estimated glomerular filtration rate | 180 days after procedure
  Secondary endpoints were the relative reduction in estimated glomerular filtration rate (eGFR) as well as all cause mortality, myocardial infarction and stent thrombosis at 30-day and 180-day after procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China